CLINICAL TRIAL: NCT06622278
Title: Flipped Classroom for Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Donnelly, Director, Division for Physical Activity and Weight Management, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCRP - S1
Record Dates: First submitted 2022-06-13; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Health Education (Experimental): Participants will be complete a total of 24, 1-hour group sessions with a health educator (exercise physiologist). The group size will be 10-15 participants and will be completed via Zoom. Prior to each group meeting, participants will email their weekly self-monitoring sheets to their health educator to review diet and exercise adherence. Each group session will follow a pre-determined structure: group discussion, review of adherence, 5 to 10 minutes of physical activity, and an active learning-based activity.
  Interventions: Behavioral: Flipped Classroom

INTERVENTIONS:
Behavioral: Flipped Classroom — The flipped classroom educational model requires participants to independently review educational material before class, and class time with the health educator is spent engaging in group and individual skills-based activities and problem-solving assignments. The theoretical basis for the development of active learning is to elicit higher cognitive learning, according to the revised Bloom's taxonomy and shift independent student time to passive learning (remembering and understanding) and collaborative student and educator time to active learning (applying, analyzing, evaluating, and creating). Thus, the weight management education will include: case vignettes, group debates/discussions, think-pair-share activities, gamification of health-related topics, creation of meal and physical activity, problem-solving barriers to a healthy diet and physical activity, and hands-on worksheets.

SUMMARY:
This study is a 24-week, single-arm trial investigating the feasibility of a flipped classroom behavioral intervention for weight management. The investigators will recruit up to 30 adults ages 18+ with a body mass index greater than or equal to 25 kg/m2 to participate in weekly, 1-hour group weight management education delivered remotely via Zoom with a trained health educator. Participants will receive a dietary prescription of 1200-1500 calories/day (5 portion-controlled meals and 5+ servings of fruits and vegetables) and exercise prescription of 150-300 minutes exercise/week. Additionally, participants will be asked to self-monitor diet and exercise adherence weekly. Feasibility outcomes will be collected at baseline, 12-weeks, and 24-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than or equal to 25
* Age 18 to 75 years
* Wireless internet connection in the home
* Ability to engage in moderate to vigorous intensity exercise

Exclusion Criteria:

* Unable to commit to weekly group education
* Food allergy/intolerance that would hinder ability to adhere to dietary prescription

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Attendance | 24 weeks
  Attendance to the group education sessions will be measured weekly and evaluated by the health educator. Attendance records will be entered into the study REDCap database.
Attrition | 24 weeks
  Attrition rate will be measured at the end of the intervention measured as the percent of participants who completed all 24 weeks of the weight loss program.

SECONDARY OUTCOMES:
Weight | 24 weeks
  Participants will be weighed at the outpatient weight management clinic in a private room by a registered nurse prior to the participant seeing a clinic physician. Weight will be collected to the nearest 0.1 kg.
Height | 24 weeks
  Participant height will be measured at the outpatient weight management clinic in a private room by a registered nurse prior to the participant seeing a clinic physician. Standing height will be measured using a stadiometer and collected to the nearest 1 cm.
Body Mass Index | 24 weeks
  Body Mass Index will be calculated as weight (kg) divided by height (cm) squared.
Diet Adherence | 24 weeks
  Adherence to the diet prescription will be measured weekly via participant self-report. Participants will report daily total number of shakes, number of entrees, servings of fruit and vegetables, and days off plan. The self-monitoring sheet will be submitted via email to the health educator prior to each group session. The health educator will provide individual feedback based on self-reported adherence.
Exercise Adherence | 24 weeks
  Adherence to the diet and exercise prescription will be measured weekly via participant self-report. Participants will report daily minutes of exercise and steps taken. The self-monitoring sheet will be submitted via email to the health educator prior to each group session. The health educator will provide individual feedback based on self-reported adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT06622278/Prot_SAP_000.pdf